CLINICAL TRIAL: NCT06404814
Title: Effectiveness of Functional Electrical Stimulation Versus Spencer Technique in Patients With Adhesive Capsulitis
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Superior University (Other)
Responsible Party: Principal Investigator, Muhammad Naveed Babur, Principal Investigator, Superior University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: MSRSW/Batch-Fall22/707
Record Dates: First submitted 2024-05-05; First posted 2024-05-08 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Adhesive Capsulitis
MeSH Terms: conditions — Bursitis | interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Transcutaneous electrical nerve stimulation (TENS) (Other)
  Interventions: Behavioral: Transcutaneous electrical nerve stimulation (TENS)
- Muscle Energt Techinique (METs) (Experimental)
  Interventions: Diagnostic Test: Muscle Energy Technique

INTERVENTIONS:
Behavioral: Transcutaneous electrical nerve stimulation (TENS) — (TENS) is a method of pain relief involving the use of a mild electrical current
  Arms: Transcutaneous electrical nerve stimulation (TENS)
Diagnostic Test: Muscle Energy Technique — n Spencer's technique, there are seven steps as follows: shoulder extension along with elbow flexion, shoulder flexion with elbow extension, circumduction with compression, circumduction with distraction, shoulder abduction and internal rotation with elbow flexion, shoulder adduction and external rotation with elbow
  Arms: Muscle Energt Techinique (METs)

SUMMARY:
This study focus on the rehabilitation of patients with frozen shoulder through a manual technique called "Spencer MET".The purpose of this approach is to reduce the pain and improve the ROM and quality of life.

DETAILED DESCRIPTION:
By comparing the effectiveness of functional electrical stimulation versus the Spencer technique in patients with adhesive capsuilitis is to determine which treatment approach will yields better outcomes in order to reduce the detrimental effects of disease process.Spencer METs consist of series of seven steps taken in order to decrease pain and stiffness in sholder regiegionn.

ELIGIBILITY:
Inclusion Criteria:

* Patients with diabetic frozen shoulder
* Patients having frozen shoulder after stroke
* Subjects having stiff shoulder for at least 3 months
* Subjects with bilateral/unilateral frozen shoulder
* Subjects with idiopathic frozen shoulder

Exclusion Criteria:

* Bone fracture within past 12 weeks
* Patients with hyper mobile joints
* Subjects with Rotator cuff pathology
* Dislocated shoulder
* Subjects who had shoulder arthroplasty

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-05-01 (Actual); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
Visual Analogue Scale (VAS): | 12 Months
  It is tool widely used to measure the intensity of pain and discomfort.VAS effectively used in randomized controlled trials for outcome measures,consisting of 10 cm straight line from 0 to 10.0 represents "No pain" and 10 represent "Worst pain". Patients can mark their severity of pain.
Goniometer | 12 months
  Goniometer is instrument used to measure the range of motion of a joint.

CONTACTS AND LOCATIONS:
Locations (1):
- Johar pain relief center, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No